CLINICAL TRIAL: NCT01170754
Title: A Prospective, Randomized Controlled Trial Comparing the Efficacy and Patient Tolerability of Miralax (PEG 3350) vs. Golytely as Bowel Preparation for Screening Colonoscopy
Brief Title: Miralax (PEG 3350) vs. Golytely as Bowel Preparation for Screening Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEG-3350
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Colon Cancer
Keywords: PEG-3350, polyethylene glycol, colonoscopy
MeSH Terms: conditions — Colonic Neoplasms | interventions — polyethylene glycol 3350; gatorade; Polyethylene Glycols; Electrolytes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-3350 and Gatorade (Experimental): 255 miralax with 64 oz gatorade.
  Interventions: Drug: PEG-3350 and Gatorade
- Golytely 4 Liters (Active Comparator): Golytely 4 Liters
  Interventions: Drug: Golytely 4 liters

INTERVENTIONS:
Drug: PEG-3350 and Gatorade — 255 grams of miralax mixed with 64 ounces gatorade for colonoscopy preparation.
  Other Names: nulytely, PEG-3350, Miralax, glycolax
  Arms: PEG-3350 and Gatorade
Drug: Golytely 4 liters — Golytely 4 liters
  Other Names: polyethylene glycol/electrolytes
  Arms: Golytely 4 Liters

SUMMARY:
A major limitation to the widespread acceptance of colonoscopy as a procedure to screen for colorectal cancer is the laxative preparation. Phosphate-based preps (e.g. Fleets Phosphosoda) are now used on a limited basis because of their known association with renal injury. Polyethylene glycol (PEG) mixed with a balanced electrolyte solution (e.g. Golytely) has been used for over two decades for colon cleansing. The mixture is not very palatable due to the electrolyte additives which include sodium sulfate.

To overcome the limitation of existing preps, gastroenterologists and colorectal surgeons worldwide have been using PEG powder alone (same quantity as found in Golytely prep) not mixed with electrolytes (Glycolax or Miralax) and dissolving this into 64 ounces of Gatorade. Conservatively, we estimate that 25% of colonoscopies in the US are being done with this prep. Anecdotally there have been reports (case series) that it is far more palatable and the prep is equally efficacious. The active ingredient, PEG, is not changed and therefore this is not surprising. The issue at present is that there has never been a blinded study to confirm these claims.

This study will compare the efficacy of the two preps. There is no funding. The investigators will charge insurance companies for the prep - this is our current practice. The procedures will be done on healthy individuals referred for colon cancer screening and the exam will be billed to their insurance. There will be no patient honorarium. The investigators will check electrolytes to be sure patients do not develop hypokalemia with the Gatorade prep.

DETAILED DESCRIPTION:
Objective To determine whether Miralax is as efficacious for bowel cleansing as standard Golytely for screening colonoscopy. This study is designed and powered to be an non-inferiority study.

Primary aim: To compare the quality of bowel preparation between Miralax and Golytely

Secondary Aims:

* compare patient comfort and tolerability with each of the 2 preparation regimens
* evaluate the effects of age, gender and tolerability on bowel prep quality
* to determine if either preparation is associated with acute electrolyte disturbances

Background Colonoscopy is the standard method for luminal evaluation of the colon. Bowel cleansing prior to colonoscopy is critical to the endoscopist obtaining optimal visualization during the procedure and therefore plays an integral role in safety, efficacy and diagnostic accuracy of the procedure. The bowel cleansing portion of the procedure is often the most lamented aspect of the colonoscopy experience. This is often driven by the large volume of liquid required to be consumed, in addition to the poor palatability of some colon cleansing regimens. Cleansing methods are variable, and often times high volume solutions are time consuming, inconvenient and uncomfortable, leading to poor patient compliance. This translates into decreased effectiveness of the colonoscopy exam and often higher costs due to the need for repeat examination. Additionally, it is unknown how much the feared discomfort of the bowel preparation experience dissuades patients from pursuing a screening colonoscopy for colon cancer.

An ideal bowel preparation would reliably cleanse the colon in a rapid fashion, would not alter the colonic mucosa, result in an acceptable amount of patient discomfort, would not cause significant shifts in electrolytes and would be inexpensive. To date, no bowel regimen meets all of these criteria.

One of the standard bowel preparation regimens is polyethylene glycol (PEG, Golytely) lavage solution which entails consuming 4 L of water mixed with a powder packet that contains the main ingredient (255g polyethylene glycol 3350) along with electrolytes (22.74 g anhydrous sodium sulfate, 6.74 g sodium bicarbonate, 5.86 g sodium chloride, 2.97 g potassium chloride). This is a non-absorbable, iso-osmotic solution which has a mildly salty taste that induces a diarrhea that rapidly cleanses the bowel, usually within 4 hours. This solution was first introduced in the 1980's and is currently the most widely used bowel cleansing regimen (1). It has proven safety and efficacy but due to its high volume, it is often difficult for patients to tolerate (2-7). It has been estimated that at least 5-15% of patients do not complete the preparation due to the large volume and/or poor palatability (8, 9). The literature also confirms that patients prefer lower volume solutions for comfort and tolerability (7, 10).

Oral sodium phosphate solutions (e.g. Fleets PhosphoSoda®) were equally efficacious and shown to be better tolerated low volume alternatives to PEG (11). They were FDA approved for bowel cleansing and were been used extensively in select patients prior to colonoscopy until recently. However, on December 11, 2008, the FDA issued a statement concluding that the use of oral sodium phosphate preparations poses a risk of serious adverse events, notably acute phosphate nephropathy- a type of acute kidney injury- in select patients (patients over age 55, baseline kidney disease, on diuretics, angiotensin converting enzyme [ACE] inhibitors, NSAIDs or angiotensin-receptor blockers [ARBs] etc) (12-14). As a result, the FDA has required that manufacturers of oral sodium phosphate bowel preparations add a Boxed Warning to their labels of these products. Subsequently, these manufacturers have voluntarily removed their products from retail sale. There have been over 20 randomized controlled trials in the literature searching for the "ideal" bowel preparation (11). With the removal of oral sodium phosphate preparations from the market, the search for a better tolerated bowel cleansing regimen continues.

Miralax (PEG 3350), polyethylene glycol powder alone without electrolytes is FDA approved for constipation. It is mixed in 8-12 ounces of any beverage and can be used daily. Because it lacks taste (no electrolytes) it has been used as a bowel cleanser for colonoscopy. Generally, 255 g of Miralax is combined with 64 oz of Gatorade for bowel cleansing prior to colonoscopy. While not FDA approved for this indication, it has been widely used and is an accepted alternative to Golytely in numerous endoscopy centers across the country.

PEG 3350's safety and efficacy has been documented in multiple studies on children undergoing colonoscopy (15, 16). A recent single arm feasibility study described in a letter to the editor in the American Journal of Gastroenterology 2008 found the use of Miralax (PEG 3350) as colonoscopic preparation to be tolerable and safe in adults (17). Moreover the study reported high compliance. It included 29 patients who underwent screening colonoscopy with PEG 3350 in 64 oz of Gatorade® (The Gatorade Company, Chicago, IL). A "good prep" was described in 97% of cases; patient rated tolerance was good in 86%. Insomnia was the most common adverse effect. Of note, 18 patients had prior 4L PEG bowel cleansing experiences- of these, 50% reported PEG 3350 was better tolerated. Beyond this data, these investigators at a community center (Urbana, IL) have a 3 year exclusive experience with PEG 3350 as their colon preparation; they report anecdotally better patient tolerance and compliance over prior preparations. The inclusion of Gatorade® is to reduce the potential for electrolyte disturbances.

In addition to its low volume, PEG 3350 (Miralax) is storied to be more palatable and easily accessible over the counter; it is also a simple, uncomplicated regimen. Based on the theory that greater ease of use, improved taste, lower volume and lower levels of induced discomfort would result in better patient compliance, completion of the bowel preparation and subsequent improvement in visualization during colonoscopy, PEG 3350 (Miralax) appears to be promising as an "ideal" cleansing agent. To date, there has been no head to head comparison of MiraLAX and Golytely in terms of efficacy and patient tolerability as bowel cleansing regimens for colonoscopy.

Eligibility Criteria Inclusion criteria

* All adults undergoing average risk colon cancer screening (ages 40-75 years old)
* Able to provide informed consent

Exclusion criteria

* A history of constipation
* Patients who use medications to assist with a bowel movement such as osmotic, stimulant, or cathartic laxatives (including "colon cleansers")
* Diabetes or glucose intolerance
* Patients with severe underlying renal or hepatic impairment
* Pregnant women - pregnancy test performed on all menstruating women before procedure.

Treatment Plan This is a prospective, randomized, endoscopist-blinded study that will be carried out at Temple University Hospital. All adult patients undergoing outpatient colonoscopy will be screened for enrollment in the study.

Upon completion of a history and physical, patients identified as appropriate for the study will be approached about study participation. Informed consent by the PI will be completed in the outpatient office and the patient will be scheduled for colonoscopy. The risks and benefits of the exam will also be discussed. Once the patient is scheduled, the medical assistant scheduling the exam will open an opaque envelope and assign the patient their exam preparation. She will give a script for Golytely or Miralax. Gatorade must be purchased by the participant. The details of the bowel preparation are below:

* All patients will be advised to have clear liquids for breakfast, lunch and dinner on the day prior to their planned colonoscopy.
* Based on their randomization assignment, subjects will be instructed to either

  1. Consume 4 L polyethylene glycol (Golytely) Or
  2. Consume 255 g of PEG 3350 (Miralax) in 64 oz of yellow Gatorade. The choices will be the Lemon-Lime , Lemonade, or All-Stars Lemon Lime flavors which are all primarily yellow.

Study participants will be instructed to take nothing by mouth after midnight on the day of their colonoscopy. They will also be advised to avoid discussing the details of their bowel preparation with their endoscopist until after their colonoscopy. Upon arrival to their scheduled colonoscopy appointment and prior to their procedure, patients will be provided a short survey assessing their bowel preparation experience (please refer to appendix document Patient Survey for details). Also at the time of insertion of an intravenous catheter (which is required for all procedures) 5 cc of blood will be drawn for a complete metabolic panel and sent to the TUH laboratory to evaluate for electrolyte disturbances.

All procedures will be performed at the Temple University Hospital Digestive Disease Center by the PI. He will be blinded to the type of bowel preparation randomized to the patient. Upon completion of the procedure, the endoscopist will document the adequacy of the preparation (24). The preparation quality will be assessed for each portion of the colon according to the following scale (see appendix):

Boston Bowel Prep Scale 0 unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared

1. portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen because of staining, residual stool and/or opaque liquid
2. minor amount of residual staining, small fragments of stool, and/or opaque liquid, but mucosa of colon segment is well seen
3. entire mucosa of colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid

A sum score will be calculated based on the rating in each colonic segment. In order to assess validity and reliability in the rating scale both intra-observer and inter-observer reliability will be assessed. This will be done by taking representative high resolution digital photographs of all colonic segments during the withdraw phase of the colonoscopy. The photographs will be printed and de-identified. At the end of the study the PI will blindly grade each prep using photographs presented in a random fashion. A second experienced colonoscopist from the Temple faculty will also grade each prep to assess inter-observer reliability.

Risks The risks of this study include the use of a colonoscopy bowel preparation agent that is not FDA approved for this indication as well as the inherent risk of colonoscopy. The added risks of this study are only related to the preparation. Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. The risks of undergoing colonoscopy include bleeding potentially requiring transfusion of blood products, infection, bowel perforation possibly requiring surgical intervention, adverse reaction to anesthesia/sedation, and missed lesions. These risks are rare and are standard for any colonoscopic exam regardless of study participation.

Benefits The benefits afforded to study subjects would include potential early detection and treatment of colorectal cancer, prevention of colorectal cancer by removal of pre-malignant polyps and development of a cancer prevention or surveillance strategy based on colonoscopic findings. Also, 50% of the patients will consume a preparation that is likely to be far more palatable than the standard preparation, Golytely.

Alternative Treatments Cancer prevention tests should be offered to all patients meeting criteria for CRC screening. The preferred cancer prevention test is colonoscopy. Alternative cancer prevention tests include flexible sigmoidoscopy and computed tomography colonography. Patients who decline colonoscopy or a cancer prevention test should be offered a cancer detection test. The preferred cancer detection test is fecal immunochemical testing. Alternative cancer detection tests included Hemoccult Sensa fecal guaiac based testing and fecal DNA testing. No CRC screening is an alternative.(1)

Data Collection and Statistics Sample Size Calculation The primary objective of the study is to compare the efficacy, tolerability and safety of the standard bowel preparation Golytely with a novel bowel preparation agent Miralax. The study is a non-inferiority study: The objective is to conclude that the prep quality scores of those receiving Miralax is at most 10% less than for Golytely. Thus the difference in prep scores between Miralax minus Golytely should be greater than - 10%. If this is the case, Miralax would be considered as non-inferior to Golytely. To calculate sample size we performed a one-sided test based on the binomial distribution with the intent of demonstrating that Miralax is non-inferior if the calculated one-sided p-value is less than 0.05. If the true difference between the Miralax and Golytely is exactly 0%, then the test should give a p-value less than 0.05 with a probability of 0.80. Since we want to conclude that the difference in responders, Miralax minus Golytely, is greater than - 10%, we choose as the null hypothesis H0: the true difference in proportions is less than or equal to - 0.10 and the alternative hypothesis H1: the true difference in proportions is greater than - 0.10. Based on the study by Lai and others (24), on a 0-9 scale the expected mean prep score with Golytely will be 6.2 with a standard deviation of 1.5.

Below is the output from PASS 2008 (Kaysville, UT ) Power Analysis of a Non-Inferiority Test of The Difference of Two Means Numeric Results for Non-Inferiority Test (H0: D <= -|E|; H1: D > -|E|)

Test Statistic: T-Test:

Power N1/N2 (E) (D) (Alpha) Beta (SD1) (SD2) 0.80019 78/78 -0.600 0.000 0.05000 0.19981 1.500 1.500 Report Definitions Group 1 is the treatment group. Group 2 is the reference or standard group. N1 is the number of subjects in the first (treatment) group. N2 is the number of subjects in the second (reference) group.

|E| is the magnitude of the margin of equivalence. It is the largest difference that is not of practical significance.

D is the mean difference at which the power is computed. D = Mean1 - Mean2. Alpha is the probability of a false-positive result. Beta is the probability of a false-negative result. SD1 and SD2 are the standard deviations of groups 1 and 2, respectively. Summary Statements Group sample sizes of 78 and 78 achieve 80% power to detect non-inferiority using a one-sided, two-sample t-test. The margin of equivalence is -0.600. The true difference between the means is assumed to be 0.000. The significance level (alpha) of the test is 0.05000. The data are drawn from populations with standard deviations of 1.500 and 1.500. Statistical Analyses Statistical analyses will be conducted by using statistical software (SPSS 17.0). The proportions in 2 x2 contingency tables will be compared by the chi square test. The investigators will use a kappa statistic to evaluate for inter-observer and intra-observer variability in the bowel preparation quality. Multivariate analysis will be performed with multiple logistic regression to assess the impact of age and gender on bowel preparation. The investigators plan to have complete follow up of all patients and will use an intention to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

All adults undergoing average risk colon cancer screening (ages 40-75 years old)

•Able to provide informed consent

Exclusion Criteria:

* A history of constipation
* Patients who use medications to assist with a bowel movement such as osmotic, stimulant, or cathartic laxatives (including "colon cleansers")
* Diabetes or glucose intolerance
* Patients with severe underlying renal or hepatic impairment
* Pregnant women - pregnancy test performed on all menstruating women before procedure.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Friedenberg, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McKenna T, Macgill A, Porat G, Friedenberg FK. Colonoscopy preparation: polyethylene glycol with Gatorade is as safe and efficacious as four liters of polyethylene glycol with balanced electrolytes. Dig Dis Sci. 2012 Dec;57(12):3098-105. doi: 10.1007/s10620-012-2266-5. Epub 2012 Jun 19. PMID 22711499

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-3350 and Gatorade: 255 miralax with 64 oz gatorade.
  Golytely vs. Miralax plus gatorade: 4L of golytely vs. 255 grams of PEG-3350 mixed with 64 ounces gatorade for colonoscopy preparation.
- Golytely 4 Liters: Golytely 4 Liters
  Golytely vs. Miralax plus gatorade: 4L of golytely vs. 255 grams of PEG-3350 mixed with 64 ounces gatorade for colonoscopy preparation.
Period: Overall Study
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Started | 66 | 70
Completed | 66 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters | Total
Number analyzed (Participants) | 66 | 70 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 64 | 124
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (8.4) | 56.7 (7.0) | 56.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 44 | 74
  Male | 36 | 26 | 62

OUTCOME MEASURES:

1. Primary Outcome: Boston Prep Scale
Description: The study is a non-inferiority study: The objective is to conclude that the prep quality scores of those receiving Miralax is at most 10% less than for Golytely. Thus the difference in prep scores between Miralax minus Golytely should be greater than - 10%. If this is the case, Miralax would be considered as non-inferior to Golytely.
  The outcome measure will use the Boston Prep Scale. The BPS is scored 0-9 with 9 being an excellent preparation throughout the colon. From the right colon, transverse colon , and left colon a score of 0-3 is given as follows and the total BPS is the arithmetic sum from each colon segment:
  0 = Unprepared colon segment with mucosa not seen due to solid stool.
  1. = Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen.
  2. = Minor amount of residual staining, small fragments of stool and/or opaque liquid
  3. = clear colon without staining
Time Frame: photographs were taken throughout the colonoscopy and reviewed within 1 month after procedure.
Population: Includes all subjects who were enrolled and underwent procedure (Intention-to-treat analysis)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
units on a scale | 7.0 (2.1) | 7.2 (1.9)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Non-Inferiority — Inferiority between the two groups was defined as a difference of 10% in the overall BBPS score; p = .45, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

2. Secondary Outcome: Sodium Level in mmol/L
Description: Sodium level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mmol/L | 138.8 (2.4) | 139.3 (2.4)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .13, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

3. Secondary Outcome: Potassium Level in mmol/L
Description: Potassium level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mmol/L | 4.0 (3.2) | 3.9 (3.5)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .31, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

4. Secondary Outcome: Chloride Level in mmol/L
Description: Chloride level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mmol/L | 104.1 (2.6) | 104.2 (3.2)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .87, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

5. Secondary Outcome: Bicarbonate Level in mmol/L
Description: Bicarbonate level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mmol/L | 26.4 (2.5) | 25.9 (2.5)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .25, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

6. Secondary Outcome: BUN Level in mg/dl
Description: BUN level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mg/dl | 9.0 (3.4) | 9.5 (4.0)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .47, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

7. Secondary Outcome: Creatinine Level in mg/dl
Description: Creatinine level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mg/dl | 0.9 (0.19) | 1.1 (2.0)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .34, t-test, 2 sided

8. Secondary Outcome: Glucose Level in mg/dl
Description: Glucose level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mg/dl | 98.2 (12.2) | 93.7 (21.5)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .18, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

9. Secondary Outcome: Calcium Level in mg/dl
Description: Calcium level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mg/dl | 9.3 (0.35) | 9.3 (0.46)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .75, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

10. Secondary Outcome: Magnesium Level in mg/dl
Description: Magnesium level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mg/dl | 2.1 (0.20) | 2.1 (0.26)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .92, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

11. Secondary Outcome: Phosphorus Level in mg/dl
Description: Phosphorus level: Risks from the preparation include failure to cleanse the colon adequately and the risk of electrolyte abnormalities, particularly hypokalemia. We will compare adverse events from the comparator preps by assessing electrolytes on the day of the procedure.
Time Frame: Day of procedure
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 66 | 70
mg/dl | 3.4 (0.52) | 3.5 (0.60)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Equivalence — Equivalence between the two groups was defined as a p-value = or >.05; p = .60, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

12. Other Pre Specified Outcome: Boston Prep Scale (Per Protocol Analysis)
Description: Analysis includes a sub-group of subjects who drank >75% of the preparation and adhered to a clear liquid diet (Per Protocol).
  The BPS is scored 0-9 with 9 being an excellent preparation throughout the colon. From the right colon, transverse colon , and left colon a score of 0-3 is given as follows and the total BPS is the arithmetic sum from each colon segment:
Time Frame: photographs were taken throughout colonoscopy and reviewed within 1 month after procedure
Population: Includes subjects who followed instructions (Per Protocol analysis)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Number analyzed (Participants) | 50 | 54
units on a scale | 7.4 (1.8) | 7.4 (1.7)
Statistical Analysis 1: Comparison: PEG-3350 and Gatorade vs Golytely 4 Liters; Test type: Non-Inferiority — Inferiority between groups was defined as a difference of 10% in the overall BBPS score; p = .98, t-test, 2 sided — p<.05 was defined as the a priori threshold for statistical significance

ADVERSE EVENTS:
Time Frame: Only for the day of the procedure for electrolytes and 24 hours later for symptoms after procedure and complications from colonoscopy.
Description: We checked a basic metabolic profile on day of colonoscopy. All patients called the day after procedure to assess for complications.
Arm/Group | PEG-3350 and Gatorade | Golytely 4 Liters
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/70
Other Adverse Events (participants affected / at risk) | 4/66 | 4/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-3350 and Gatorade (N=66) | Golytely 4 Liters (N=70)
Hypokalemia (Renal and urinary disorders) | 4 (4) | 4 (4) — These adverse events were for potassium levels between 3.0-3.5 meq/ml.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No